CLINICAL TRIAL: NCT06506162
Title: The Effect of Flavor and Nicotine Strength on the Abuse Liability and Appeal of Oral Nicotine Products
Brief Title: Abuse Liability and Appeal of Oral Nicotine Products
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Robert Monterosso, Assoc Prof Psychology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UP-22-00228; U54CA180905 (NIH)
Record Dates: First submitted 2024-07-03; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Flavoring Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Nicotine Gum (Active Comparator): Participants in this arm will only use Lucy brand 2mg nicotine gum
  Interventions: Other: Flavor; Other: Nicotine concentration
- High Nicotine Gum (Active Comparator): Participants in this arm will only use Lucy brand 6mg nicotine gum
  Interventions: Other: Flavor; Other: Nicotine concentration
- Low Nicotine Pouch (Active Comparator): Participants in this arm will only use ON! brand 2mg nicotine pouches
  Interventions: Other: Flavor; Other: Nicotine concentration
- High Nicotine Pouch (Active Comparator): Participants in this arm will only use ON! brand 6mg nicotine pouches
  Interventions: Other: Flavor; Other: Nicotine concentration

INTERVENTIONS:
Other: Flavor — The study will compare sweet vs. cool flavors
Other: Nicotine concentration — The study will compare low vs. high strength Oral Nicotine Products

SUMMARY:
There has been a recent proliferation of novel oral nicotine products (ONPs) brought to market, including new nicotine gums and pouches. Unlike electronic cigarettes (ECs) ONPs have no impending regulatory barriers with regard to flavoring or nicotine dose, and manufacturers have capitalized on this by introducing an extensive slate of characterizing flavors and nicotine concentrations. Both sales trajectory and the surge in marketing suggest ONP use is likely to increase in the coming years. Work by the investigators and others indicates that interest in these products is high among current EC users, and among specific demographic groups including those who identify as sexual and gender minority (SGM). ONP use is discrete and so can function as a secondary source of nicotine, encouraging dual use patterns and more severe nicotine dependence. Depending on the use patterns of ONPs that emerge, regulation of ONPs may serve the public health interest. However, very little is known about factors relevant to the actual appeal and abuse liability of these products. The investigators propose to address this important gap by assessing the appeal and abuse liability of gum and pouch ONPs as a function of flavor (mint vs fruit) and nicotine concentration (2mg vs. 4mg). Flavor and nicotine strength, along with product type, are regulatable attributes, and so it is essential to understand their impact on appeal and abuse liability. Evidence from EC use suggests a potential interaction between flavor and nicotine strength, with flavorants in the "mint" category desensitizing receptors integral to the aversive sensory experience of nicotine, leading to greater tolerability of high nicotine concentration. Because of current ONP marketing emphasis on youth, the investigators will recruit young adult exclusive EC users (N = 320; ages 21 - 25). The investigators will target recruitment of a sufficient number of SGM participants (N = 64, 20% of sample) to allow assessment of potential differentiation of this group. Participants will complete one virtual session focused on assessment of the sensory appeal of ONPs. Based on individual participant ratings, the preferred fruit and the preferred mint ONP will be selected (from their randomized product type and nicotine strength) to each be assessed in a single-product session examining factors known to predict abuse liability (relief of withdrawal, liking, behavioral economic indices of demand, and follow-up naturalistic product use). The investigators will pay particular attention to evidence suggesting dual use potential of ONPs, given its association with greater severity of nicotine dependence. The proposed work will inform efforts to mitigate ONPs potential to promote dual-use and more severe nicotine dependence among young adult EC users, by isolating the impact of potential regulatory targets.

DETAILED DESCRIPTION:
E-cigarettes (ECs) have been the predominant flavored non-combustible tobacco product used by young adults since 2014,(Ali et al. 2022) and are disproportionately used by sexual/gender minorities (SGM) (Buchting et al. 2017;Wheldon et al. 2019)). However, patterns are likely to change due to: 1) increasing regulatory restrictions on non-tobacco flavored ECs, and 2) the emergence new nonmedicinal oral nicotine products (ONPs; e.g., pouches and gums) with enhanced palatability (e.g., improved flavoring) (Lunell et al. 2022). Preliminary data shows that many young adult e-cigarette users with no intention to quit vaping perceive ONPs as secondary means of nicotine consumption when vaping is prohibited. Because EC+ONP dual use could exacerbate nicotine dependence by increasing daily nicotine intake, it is important to identify drivers of ONP appeal and abuse liability in young adult EC users to inform regulations that prevent adverse dual use in young people. Nicotine concentration and flavors are two putative drivers of ONP appeal and abuse liability, given that ONPs deliver substantial buccal nicotine absorption(Lunell et al. 2022) and, like ECs, their flavors elicit pleasant sensory effects (Goldenson et al. 2019; Leventhal et al. 2020). Certain ONP flavors may offset nicotine's oral irritating effects via anesthetizing cooling effects (mint flavored ONPs with menthol), allowing tolerability of higher doses of nicotine. ONP type may also be important to ONP appeal. Initial evidence (primarily product interest survey data) suggests young adult EC users and adolescents may have higher affinity for nicotine gum than pouches, and interest in using ONPs was greater within certain vulnerable populations, especially SGMs.

The investigators will determine the appeal and abuse (including dual use) liability of gum and pouch ONPs as a function of flavor (mint vs fruit) and nicotine concentration (gum 2mg vs. 6mg; pouch 2mg vs. 6mg) among young adult exclusive EC users (N = 320; ages 21 - 25). Data will be collected via virtual study sessions in which participants residences become 'remote laboratories' (allowing nationwide quota sampling). Following an orientation, participants will be randomized to one of two ONP types (gum or pouch) and nicotine concentrations (low vs. high), resulting in four study groups. The randomized nicotine-ONP combination will then be tested in: (i) a single-visit appeal/sensory attribute testing involving controlled self-administration of mint and fruit flavored ONPs; and (ii) two abuse liability evaluations (one for fruit one for mint) each involving a single-visit controlled ONP self-administration session and 1-week post-visit naturalistic use of the respective ONP.

Overview of Project. The investigators will utilize an experimental design to determine the acute appeal and abuse liability of gum and pouch ONPs among young adult current EC users. Data will be collected via three online sessions with participants from across the US in which their own residences become a 'remote lab.' Following an orientation session, participants will be randomized to one of four groups varied by product type ( a gum or pouch) and nicotine concentration (low [2mg] or high [6mg]) and receive that type and nicotine level throughout the entire protocol. Experimental session 1 (Sensory Appeal session) collect ratings appeal and sensory attributes directly after self-administering 2 fruit (e.g., citrus, pomegranate) and 2 mint (e.g., spearmint, wintergreen) flavored variants of their ONP type/nicotine condition in in a single visit. Order of the 4 flavors will be in one of 24 possible sequences randomly assigned for each participant. The highest rated fruit variant and highest rated mint variant will be selected for the subsequent two sessions. Experimental sessions 2 & 3 (Abuse Liability sessions) involve 30-min self-administration of one ONP (fruit ONP in one session, mint ONP in another session; order counterbalanced) in separate sessions after 18-hours of abstinence. Dependent variables will include withdrawal/urge suppression, subjective effects, and behavioral economic indicators of reward value. In addition, for the 7 days after each abuse liability session visit participants will report on naturalistic use of the same product (a free provision of 30 pieces of each product that was administered in the previous Abuse Liability session will be provided to participants to use ad lib).

Rationale for Methods. (Overall design rationale) Rationale for the two-part appeal + abuse liability protocol: Based on the integration of paradigms that the investigators developed to assess abuse liability and appeal of ECs, a two-part protocol will be used. The first experimental session (Sensory Appeal session) in the proposed design provides information about the sensory attributes of the user experience that drives appeal of different flavors. Given that multiple products (four) are tested within a single visit, and appeal ratings are collected immediately during use, differences across flavors are driven by sensory experience and cannot be attributed to differences driven by the neuropharmacological effects of nicotine. By contrast, the Abuse Liability experimental sessions (Sessions 2 - 3) test a single flavored product within a session, which will provide a richer source of information about the use and valuation of ONPs due to the combination of the sensory and neuropharmacological effects.

Justification of mixed factorial design. While a fully within-participant design would provide the greatest power to detect divergence between product conditions, an 8 multi-hour abuse liability study sessions would be too burdensome and monotonous to maintain consistent participant engagement. A mixed-factorial design allows sufficient statistical power to estimate the impact of study variables without overburdening participants.

Justification of 7-day monitoring period. Given the limited surveillance (i.e., only nicotine pouches assessed in NYTS, no measures of new ONPs in PATH or NSDUH) of these new nonmedicinal ONPs, and to better understand how young adults may use these products in conjunction with their EC, the investigators include brief (approximately 2 minutes) daily surveys assessing ONP use and use in situations when vaping is constrained. This will provide much needed data on the dual use liability of ONPs and ECs in the natural ecology, and allow assessment of whether use varies by ONP type, flavor, and nicotine strength. The investigators are well versed in utilizing remote monitoring periods to examine naturalistic use patterns of EC and polytobacco product use behaviors among young adults.

Rationale for product type and characteristics. Justification of flavors. The investigators could have focused on a particular flavoring constituent (e.g., menthol, vanillin) and designed a study around manipulating the presence or concentration of that constituent to isolate their effect. However, more than 120 different flavoring constituents have been identified in ONPs, including up to 25 flavoring constituents within a single characterizing flavor (e.g., berry) that combine to create the sensory profile. Hence, disaggregating particular constituents would not be representative of the ONP characterizing flavors sold on the market, and FDA has historically regulated according to the characterizing flavor rather than particular constituents. The TCORS methods core will do a flavoring constituent analysis which will provide contextual data on this issue. Among the characterizing flavors, the investigators focus on fruit and mint because they are the preferred EC flavor categories among AYAs and tobacco naïve individuals,(King et al. 2018) and survey data suggesting interest in ONPs of these flavors is high (see above).

Justification of nicotine concentrations. The investigators include 2mg vs. 6mg nicotine because of the prominence of these concentrations on the ONP market. However, there are ONPs currently available with substantially higher nicotine concentration (>20mg). While many ONP users report titrating up their ONP dose after they become accustomed to the sensations of ONP use, most find nicotine's irritating oral effects as uncomfortable at first. Because study participants are ONP-naïve starting with these two doses (which are low and moderate range) is indicated. The investigators also considered the inclusion of matched products without nicotine. However, the absence of any such marketed products would require imperfectly matched alternatives (e.g., confectionery gums) and would not usefully advance the primary aim of providing information directly relevant to FDA decision-making because FDA-CTP does not regulate such products.

Justification of ONP types. The investigators selected nicotine gum and pouch because extensive industry marketing is currently being directed at both products. The Center includes monitoring of additional nicotine products (including lozenges) and if they emerge as highly popular, the investigators will add lab assessments through the Center's CEC/RRP mechanism.

Eligibility, (see inclusion/exclusion section)

Procedures

Initial screening. Advertisements will phone numbers for Research Assistants (RAs), a QR code, and a direct link to an online study screener. Potentially eligible participants are contacted by RAs to conduct a detailed phone screen to confirm all self-report eligibility criteria. Eligible participants will be scheduled orientation session to be conducted over Zoom to provide informed consent.

Orientation (Consent) Session. Before the orientation, participants will be mailed supplies, including for collecting a baseline urine test of recent nicotine use involving a test strips that provide semi-quantitative total nicotine equivalents (TNEs) estimates of nicotine and nicotine metabolites (0-14 levels; >1 required for eligibility). At the outset of the orientation, presence of a computer, laptop, tablet, or similar device with working camera, microphone, and audio and Internet to complete REDCap surveys will be confirmed. After confirming age and obtaining digital informed consent, the urine nicotine test will be collected and (if positive), participants will be asked to assure that the study products shipped to participants will be kept in a safe place away from children, animals, and minors and used only for the research study. Next, self-report measures of demographics and tobacco product use history will be completed. Finally, participants will be scheduled for their next experimental visits and remined that 18-hour nicotine abstinence is required and will be confirmed by urine for each visit. To provide some control over daily fluctuations in nicotine craving and withdrawal and to facilitate adherence to the abstinence requirement, efforts will be made to complete those study visits for which abstinence is required in the morning hours (∼8:00-11:00 AM), near waking time.

Randomization to ONP type and nicotine. Participants will be randomized into one product condition (gum or pouch) and one nicotine level (high or low) stratified by region (South, West, Midwest, Northeast) and SGM status, which will determine the products used for the next 3 visits.

Provision of Appeal Session Study Materials. The investigators will mail participants a package that will include ONP products "blinded" (i.e., randomized products will be placed in labeled baggies with numbers indicating each product), remote exhaled carbon monoxide (eCO; Covita) device for biochemical verification of no combustible tobacco use, urine nicotine sample and test strip, and pregnancy test (as appropriate), product disposal bag with tamper seal tape, cleaning supplies, and materials for returning salivary samples. The eCo device is a remote device that connects to the participants cell phone device (both android and iOS) and allows for remote bioverification of smoking status (see D.5.e for cut off eCO values). The investigators will follow all safety hazard protections for product transport guidelines by shipping and courier agencies. Because this study does not involve sales of tobacco products and the products are provided for research use only, it is exempt from FDA regulations that apply to transporting tobacco products for business purposes. Study RAs will track package during shipping and inform the participant of any updates (i.e., delays, estimated arrival etc.) via phone/text. As in prior research, all sample products will be clearly labeled, "CONTAINS TOBACCO PRODUCTS, TO BE RECEIVED AND USED BY PERSON 21 YEARS OF AGE OR OLDER. FOR RESEARCH USE ONLY, NOT FOR PERSONAL USE." Upon receipt of study materials, the study team will contact the participant within 48 hours to schedule the first experimental session. In the investigators prior research providing various EC products (N = 439 experimental sessions), no study packages were opened prior to experimental sessions.

ONP Appeal Session. After confirming nicotine deprivation (semi quantitative reduction by >1 level of TNE and breath eCO of >4ppm), participants will be administered the appeal test procedure with 4 different ONPs (2 mint, 2 fruit) in random order as in prior work (e.g., Leventhal et al. 2020). Each ONP trial involves 5-minute administration period in which the product is put into the mouth (chewed [gum only] and parked between the lip and gum, per package instructions), followed by a 2-minute rating period (rate appeal and sensory attributes; see outcome measures below) and then a 2-minute water mouth rinse inter-trial interval. All products will be labeled with a letter and no identifying information about the flavor of the product will be provided to participants (i.e., participant is blinded). Prior to administration of the first product, participants will be shown a video demonstrating administration procedures. This study design has been piloted by the investigators with ONPs and was successfully implemented with ECs (over 20 ECs solutions provided and rated for appeal/sensory characteristics) in over 400 remote sessions with no adverse events.

Provision of Abuse Liability Session Study Materials. Each package will include 31 pieces/pouches of participant's top-rated fruit or mint ONPs (i.e., flavor variant with the highest appeal composite score; see below). New salivary nicotine collection kits, urine cups and pregnancy test (as appropriate), and other study materials (e.g., product disposal bag with tamper seal tape, cleaning supplies, return materials for salivary samples.

Experimental Sessions (Study Visits 2 - 3). Participants will complete two separate single-product abuse liability sessions, (one fruit, one mint; order counterbalanced across participants. After confirmand nicotine deprivation (by urine TNE and eCO). Next, pre-ONP administration withdrawal and urges will be assessed. Participants will then use the session's ONP for 30-minutes, according to a structured protocol adapted from Houtsmuller et al. (2001) for therapeutic nicotine. In this, the participant is informed to keep the ONP in their mouth for the entire 30 min. As in the previous session(s) following the chew (gum only) and park procedures, while being encouraged to move the ONP around in their mouth to where it is most comfortable. Next (post-administration phase), participants will complete withdrawal and urge follow-up measures and other questionnaires to assess specific domains relevant to abuse liability (see description below). Naturalistic 7-Day Monitoring Period: Finally, at the end of the session participants will be instructed that they may use as few or as many of the provided pieces of the session ONP over the next 7 days (30 pieces max provided to participants). Participants will report on any use through daily electronic surveys assessing frequency (e.g., number of pieces per day)/quantity (e.g., total pieces used during the monitoring period)/location of use (e.g., vape free locations, when EC is unavailable). One specific question will ask "How many times did you use the ONP in places where you normally couldn't or wouldn't vape, such as at work, indoor, or in other "smoke/vape free" locations?".

Measures. Orientation measures. Participant characteristics (demographics, vaping history (Leventhal et al. 2019), smoking history (Leventhal et al. 2019), vaping dependence (Tackett et al. 2021) flavors preferred, etc. per PhenX Toolkit) will be assessed during orientation session. Measure updates needed due to market changes (e.g., new types of flavors) will be added and developed per the MMC.

Appeal and Sensory Ratings. The investigators will use the Appeal and Sensory Quality Measures as used in Drs. Leventhal, and Monterosso's current paradigms assessing appeal and sensory attributes of ECs. Participants will rate the product on visual analog scales (range, 0-100) with answers to the following 3 questions for appeal and 4 questions for sensory attributes: (1) "How much did you like the [ONP]?"; (2) "How much did you dislike the [ONP]?"; (3) "Would you use this [product] again?"; (4) "How sweet was the [ONP]?"; (5) How bitter was the [ONP]? (6) "How much did you like the mouth feel of the [ONP]?"; 7) "How irritating or painful was the [ONP] in your mouth?". Rating anchors include "not at all" and "extremely" for each measure, except use again ("not at all" and "definitely"). The ratings of liking, disliking (reverse-scored), and willingness to use again represent related but nonredundant measures of appeal. Thus, an appeal composite score will be based on the mean of these 3 ratings per prior work (e.g., Leventhal et al., 2019). Sensory ratings will be analyze separately per previous factor analyses of ratings from EC appeal studies indicating that appeal items shared a common factor, whereas sensory attributes loaded onto distinct item-specific factors.

Abuse and Dual Use Liability. All items will be adapted for ONP language (i.e., replace vaping/smoking with ONP descriptors). Withdrawal/urge suppression (pre and post admin) Nicotine Withdrawal Scale (NWS). Nicotine withdrawal will using a validated 8-item version of the Nicotine Withdrawal Scale assessing anger/irritability, anxiety, depressed mood, restlessness/difficulty concentrating, increased appetite rated experienced right now on a scale of 0 (none/not at all) - 4 (severe/extremely) and summed. Brief Questionnaire of Vaping Urges (QVU-Brief) (Cox et al., 2001). The QVU-brief is a 10-item self-report measure with items rated from 1 (strongly disagree) to 7 (strongly agree) right now which is administered pre and post administration and yields a sum composite score. Subjective effects (post admin). Drug Effects Questionnaire (DEQ) (Morean et al., 2019). A modified version of the DEQ will be used to rate acute responses to the ONP on visual analog scales (range, 0 "not at all" - 100 "extremely"). Items assess liking/wanting (the average of "I feel good effects from the [ONP]," "I want more of that [ONP] I received," "I feel the [ONP] strength," and "I like the [ONP] effect").

The ONP Purchase Task (Cassidy et al., 2020) will assess self-reported economic demand in ONP units (gum pieces or pouches). Following a previously validated protocol (used in the investigators pilot study) purchase tasks will be completed for the ONP provided during that visit. Participants will indicate the amount of the product they would purchase for consumption for a "typical day" with no opportunity to save anything not consumed) at a series of per-unit price points. Following Mackillop et al 2008113 the following unit price points will be included: $0, $.01, $.05, $.13, $.25, $1, $2, $3, $4, $5, $6, $11, $35, $70, $140, $280, $560, and $1120. They will complete this task under two scenarios complete two hypothetical scenarios (1) Other nicotine constrained, when they are involved with no other accessible nicotine products; and (2) Vaping unconstrained the alternative specification that they have free ($0; i.e., no cost to use) access to their preferred vape. Participants will be instructed to imagine a typical day, which may or may not include periods in which vaping is prohibited or uncomfortable. Outcomes: Four measures will be derived from each task condition: Omax (the maximum total expenditure on the substance), Pmax (the price at which expenditure was highest), "intensity" (consumption at $0), and demand elasticity (a derived measure indicating the steepness with which demand drops as a function of price). Elasticity will be estimated following Hursh and Silberberg 2008,114 by fitting the demand function logQ = logQ0 + k(e-aPs - 1) where Q0 is the quantity "purchased" at $0, Ps is price if demand did not change from Q0, k is a constant across participants based on best fit to average consumption, and a is an individualized fit-parameter capturing sensitivity to price (elasticity). Since intensity, Omax, and elasticity were observed to be most predictive of nicotine use and dependence in a recent meta-analysis (González-Roz et al., 2019), these will be considered the primary three indices of demand. Dual use liability. Dual Use Liability Questionnaire (DULQ). Participants are instructed to consider times in which they want to vape but are somewhere that they don't feel they can," "To what degree is the [ONP you used today] an appealing alternative to use during those periods?", and "How willing would you be to try [the ONP] in a situation when you couldn't vape?" (a mean score of 0-7 'not at all' to 'frequently' is computed). The ONP purchase task unconstrained vs. constrained difference. Omax , Pmax , intensity, and demand elasticity will be subtracted from the respective values of the constrained variant to provide an index of dual use reward value.

Naturalistic monitoring period. Naturalistic use of provided ONPs (30 pieces/participant; ~4 pieces available/day) over the 7 days will be conducted following each Abuse Liability Session, with a brief daily survey asking how many pieces they used that day and how many pieces they have left by counting, and whether or not they used at a vape free location indoors or because they wanted to conceal nicotine use due to social concerns. Overall self-administration is assessed by the total number of pieces/pouches used (range: 0-30). Dual use self-administration. the number of days out of the week in which they reported using the ONP in a time that they felt vaping was constrained due to social concerns or indoor restrictions (0-7).

Data Analysis Plan. Data analyses will be carried out by the Center's Data Processing and Analysis Core (DPAC). The main research questions from the three Aims in the proposed study have the same structure for data analysis. Prior to primary analyses, the investigators will examine whether baseline characteristics (e.g., nicotine dependence severity, demographics) differ between the four study groups. Any sample characteristics that do differ significantly between randomized groups will be included in statistical models of study outcomes. All relevant outcome variables will be first examined with exploratory/descriptive statistical analyses that focus on describing and understanding patterns and distributions for all relevant measures (e.g., appeal ratings, desire to use again).

ELIGIBILITY:
Inclusion Criteria:

1. aged 21-25 years
2. current exclusive EC user (defined as at least weekly use over the past 3 months) and recent nicotine use confirmed by positive urine test (>1 semiquantitative Total Nicotine Equivalent; see below)
3. not currently using another tobacco/nicotine product (defined as no use in the past 6 months)
4. have never used any ONP (medicinal or nonmedicinal)
5. willing to try study provided ONPs.

Exclusion Criteria:

1. recent COVID-19+ (positive test in the past 30 days)
2. a recent COVID-19 hospitalization (past 3 months)
3. unstable or significant psychiatric conditions (past and stable conditions allowed)
4. history of cardiac event or distress within the past 3 months
5. currently pregnant (based on urine pregnancy test), planning to become pregnant, or breastfeeding.

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2028-02-14 (Estimated)

PRIMARY OUTCOMES:
Product appeal ratings | immediately after the intervention
  Participants will rate the sensory appeal of products and their motivation to use the products
Product consumption | immediately after the intervention
  Participants will have periods in which ad lib use of the product ("use as much or as little as you like") and the total used will be recorded

SECONDARY OUTCOMES:
Behavioral economic measures related to abuse liability | immediately after the intervention
  Participants will complete a purchase task that is directed at assessing valuation in the context in which alternative sources of nicotine are present, as well as when alternative sources are not present
ad lib use at home | 7 days after each abuse liability session
  participants will also receive 30 ONPs that they are free to consume during a 7 day period, with use reported each morning for the previous day

CONTACTS AND LOCATIONS:
Overall Officials: John R Monterosso, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
This study is part of the USC Tobacco Center of Regulatory Science (TCORS). We will approach data sharing in two ways: 1) USC TCORS website will include a listing of all data sets and associated data dictionaries; and 2) a formal policy will be developed for collaborative data sharing with investigators from other TCORS or other research entities. USC TCORS will provide ongoing documentation of data sets so that potential collaborators can identify opportunities to engage with the USC team and it will describe NIH policies related to collaboration and data sharing with other academics and the community. After projects have been completed and data analyzed and reported, targeting one year after completion of data collection, we will make de-identified data available generally. We will incorporate appropriate language about provision of data access into our consent processes. We will make available data codebooks, survey platforms and experimental protocols.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available within a target of 1 year after study completion
Access Criteria: To be determined

REFERENCES:
- [Background] Ali FRM, Vallone D, Seaman EL, Cordova J, Diaz MC, Tynan MA, Trivers KF, King BA. Evaluation of Statewide Restrictions on Flavored e-Cigarette Sales in the US From 2014 to 2020. JAMA Netw Open. 2022 Feb 1;5(2):e2147813. doi: 10.1001/jamanetworkopen.2021.47813. PMID 35142832
- [Background] Buchting FO, Emory KT, Scout, Kim Y, Fagan P, Vera LE, Emery S. Transgender Use of Cigarettes, Cigars, and E-Cigarettes in a National Study. Am J Prev Med. 2017 Jul;53(1):e1-e7. doi: 10.1016/j.amepre.2016.11.022. Epub 2017 Jan 13. PMID 28094133
- [Background] Wheldon CW, Wiseman KP. Tobacco Use Among Transgender and Gender Non-conforming Adults in the United States. Tob Use Insights. 2019 May 23;12:1179173X19849419. doi: 10.1177/1179173X19849419. eCollection 2019. PMID 31205426
- [Background] Lunell E, Fagerstrom K, Hughes J, Pendrill R. Pharmacokinetic Comparison of a Novel Non-tobacco-Based Nicotine Pouch (ZYN) With Conventional, Tobacco-Based Swedish Snus and American Moist Snuff. Nicotine Tob Res. 2020 Oct 8;22(10):1757-1763. doi: 10.1093/ntr/ntaa068. PMID 32319528
- [Background] Leventhal AM, Goldenson NI, Barrington-Trimis JL, Pang RD, Kirkpatrick MG. Effects of non-tobacco flavors and nicotine on e-cigarette product appeal among young adult never, former, and current smokers. Drug Alcohol Depend. 2019 Oct 1;203:99-106. doi: 10.1016/j.drugalcdep.2019.05.020. Epub 2019 Aug 1. PMID 31434028
- [Background] Goldenson NI, Leventhal AM, Simpson KA, Barrington-Trimis JL. A Review of the Use and Appeal of Flavored Electronic Cigarettes. Curr Addict Rep. 2019 Jun;6(2):98-113. doi: 10.1007/s40429-019-00244-4. Epub 2019 May 17. PMID 31453046
- [Background] Leventhal A, Cho J, Barrington-Trimis J, Pang R, Schiff S, Kirkpatrick M. Sensory attributes of e-cigarette flavours and nicotine as mediators of interproduct differences in appeal among young adults. Tob Control. 2020 Nov;29(6):679-686. doi: 10.1136/tobaccocontrol-2019-055172. Epub 2019 Dec 18. PMID 31852818
- [Background] Houtsmuller EJ, Fant RV, Eissenberg TE, Henningfield JE, Stitzer ML. Flavor improvement does not increase abuse liability of nicotine chewing gum. Pharmacol Biochem Behav. 2002 Jun;72(3):559-68. doi: 10.1016/s0091-3057(02)00723-2. PMID 12175452
- [Background] King JL, Reboussin D, Cornacchione Ross J, Wiseman KD, Wagoner KG, Sutfin EL. Polytobacco Use Among a Nationally Representative Sample of Adolescent and Young Adult E-Cigarette Users. J Adolesc Health. 2018 Oct;63(4):407-412. doi: 10.1016/j.jadohealth.2018.04.010. Epub 2018 Aug 13. PMID 30115508
- [Background] Tackett AP, Hebert ET, Smith CE, Wallace SW, Barrington-Trimis JL, Norris JE, Lechner WV, Stevens EM, Wagener TL. Youth use of e-cigarettes: Does dependence vary by device type? Addict Behav. 2021 Aug;119:106918. doi: 10.1016/j.addbeh.2021.106918. Epub 2021 Mar 23. PMID 33798918
- [Background] Morean ME, Krishnan-Sarin S, Sussman S, Foulds J, Fishbein H, Grana R, Halpern-Felsher B, Kim H, Weaver SR, O'Malley SS. Development and psychometric validation of a novel measure of sensory expectancies associated with E-cigarette use. Addict Behav. 2019 Apr;91:208-215. doi: 10.1016/j.addbeh.2018.08.031. Epub 2018 Aug 31. PMID 30197032
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Background] Cassidy RN, Long V, Tidey JW, Colby SM. Validation of an E-cigarette Purchase Task in Advanced Generation Device Users. Nicotine Tob Res. 2020 Oct 8;22(10):1851-1859. doi: 10.1093/ntr/ntaa060. PMID 32267947
- [Background] Mackillop J, Murphy JG, Tidey JW, Kahler CW, Ray LA, Bickel WK. Latent structure of facets of alcohol reinforcement from a behavioral economic demand curve. Psychopharmacology (Berl). 2009 Mar;203(1):33-40. doi: 10.1007/s00213-008-1367-5. Epub 2008 Oct 17. PMID 18925387
- [Background] Hursh SR, Silberberg A. Economic demand and essential value. Psychol Rev. 2008 Jan;115(1):186-98. doi: 10.1037/0033-295X.115.1.186. PMID 18211190
- [Background] Gonzalez-Roz A, Jackson J, Murphy C, Rohsenow DJ, MacKillop J. Behavioral economic tobacco demand in relation to cigarette consumption and nicotine dependence: a meta-analysis of cross-sectional relationships. Addiction. 2019 Nov;114(11):1926-1940. doi: 10.1111/add.14736. Epub 2019 Aug 18. PMID 31313403